CLINICAL TRIAL: NCT00578240
Title: Molecular Studies and Clinical Correlations in Human Prostatic Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Rockefeller University (Other); Flinders Medical Centre (Other Government); University of Southern California (Other); Gen-Probe, Incorporated (Industry); Genentech, Inc. (Industry); General Electric (Industry); Purdue University (Other); Biocept, Inc. (Industry); Duke University (Other); Ikonysis (Industry); Array Genomics (Industry); Cold Spring Harbor Laboratory (Other); Nodality (Industry); Epic Sciences (Industry); Rutgers Cancer Institute of New Jersey (Other); Dana-Farber Cancer Institute (Other); Johns Hopkins University (Other); M.D. Anderson Cancer Center (Other); Oregon Health and Science University (Other); University of California, San Francisco (Other); University of Chicago (Other); University of Michigan (Other); University of Washington (Other); University of Wisconsin, Madison (Other); Fred Hutchinson Cancer Center (Other); Broad Institute of MIT and Harvard (Other); Weill Medical College of Cornell University (Other); Institute of Cancer Research, United Kingdom (Other); Vitatex Inc. (Industry); Serametrix Corporation (Industry); Promega Corporation (Industry); Creatv Microtech, Inc. (Other); Viatar LLC (Industry); Massachusetts Institute of Technology (Other); Advanced Cell Diagnostics (Industry); ApoCell, Inc. (Industry); Beckman Coulter GmbH (Industry); Bioview, Inc. (Industry); Clearbridge BioMedics Pte Ltd., Singapore (Industry); Cynvenio Biosystems (Industry); Exosome Diagnostics, Inc. (Industry); Fluxion Biosciences (Industry); Foundation Medicine (Industry); Universitätsklinikum Hamburg-Eppendorf (Other); Brooklyn ImmunoTherapeutics, LLC (Industry); Ohio State University (Other); Palo Alto Research Center (Other); Rarecells (Industry); Silicon Biosystems (Industry); The Scripps Research Institute (Other); University of Minnesota (Other); Janssen Diagnostics, LLC (Industry); University of Regensburg (Other); Innocrin Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 90-040
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: benign; Rising PSA; Clinical Metastases; 90-040
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Human tissue, body fluids, and blood Fresh tissue will be obtained from patients undergoing a biopsy or surgical procedure as part of their standard therapy or as part of an investigational research protocol. Previously stored pathology specimens may also be used. Peripheral blood, bone marrow, urine, and other bodily fluids and samples will also be obtained as needed.

SUMMARY:
The Genitourinary Oncology/Urology Services at Memorial Sloan-Kettering Cancer Center (MSKCC) participates in research for the control, treatment, and cure of cancer. The purpose of this study is to collect normal and cancerous tissues, in addition to blood, and other body fluid samples from men with prostate cancer or prostatic disease. These samples may be stored for future use or used immediately by researchers who study prostate cancer and try to find better ways to diagnose, prevent, and treat it. We will look for genetic changes and protein markers on these cells. We hope to learn more about what makes some people get prostate cancer, why some cancers are more aggressive than others, and why some cancers respond to or resist different treatments. We may also try to grow the tumor cells in the lab. We may find a new treatment for prostate cancer based on this research.

DETAILED DESCRIPTION:
The therapeutics program for advanced prostate cancer is based on the hypothesis that the factors contributing to and associated with progression change as the disease evolves. To categorize these changes we now consider the disease as a series of states. 1 The states represent points where an intervention might be considered to prevent cancer from developing, to eliminate established disease, or to delay progression. The states also represent clinically significant milestones that can be used to assess treatment effects.

ELIGIBILITY:
Inclusion Criteria:

Men with prostate conditions representing the following disease states:

* No Cancer Diagnosis
* Clinically Localized Disease
* Rising PSA
* Clinical Metastases: Noncastrate
* Clinical Metastases: Castrate (Testosterone ≤ 50 ng/ml)
* Signed informed consent

Exclusion Criteria:

-Patients without any prostate related problems.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients meeting the eligibility criteria and receiving or seeking prostate cancer treatment in the Genitourinary Oncology/Urology Services will be approached by a consenting professional at a suitable point in their clinical course prior to biospecimen collection.
Sampling Method: Non-Probability Sample
Enrollment: 5290 (Actual)
Dates: Start 1990-04; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org